CLINICAL TRIAL: NCT03694717
Title: Time Course Evolution of Cardiac Output in Critically Ill Patients After a Fluid Expansion
Brief Title: Time Course Evolution of Cardiac Output
Acronym: TCCO
Status: Completed | Type: Observational
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: ADOREPS
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Acute Circulatory Failure
Keywords: shock; fluid expansion; fluid responsiveness
MeSH Terms: conditions — Shock | interventions — Saline Solution; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: The patients will receive a 500 ml fluid expansion over a standardized 10 minutes period
  Interventions: Drug: Saline Solution for Injection

INTERVENTIONS:
Drug: Saline Solution for Injection — The fluid expansion will consist in a less than 10 min infusion of 500 milliliters of saline through a central venous catheter (jugular). The duration of infusion will be controlled by an airbag pressurized at 300 mmHg.

SUMMARY:
Fluid expansion is the first therapeutic option in patients presenting acute circulatory failure but the duration of its hemodynamic effects (persistency and time of maximal increase in cardiac output) is unknown.

This study is seeking to describe in critically ill patients, the time course evolution of cardiac output over a 2-hours period after a fluid expansion.

The objectives are:

1. to identify patterns of fluid responsiveness
2. to determine the time when the maximal increase in cardiac output occurs during and a after fluid expansion
3. to compare patients' characteristics between patterns

Patients with acute circulatory failure will be recruited as soon as a fluid expansion will be decided by the physician in charge and the effects of fluid expansion on hemodynamic indices (cardiac output, arterial pressure) will be continuously recorded through a transpulmonary thermodilution device over a 2-hours period.

No changes in ventilatory settings nor vasopressors or sedatives will be allowed during the study.

Patients will be categorized into patterns according to the changes in cardiac output after fluid expansion and their characteristics will be compared.

DETAILED DESCRIPTION:
The study will be conducted in four medico-surgical ICUs in France between April 2016 and April 2018.

Since fluid challenge and invasive monitoring by thermodilution device is standard of care for septic shock management, the institutional review board waived patient consent. All patients and/or their next of kind will receive written information.

Eligible patients will have to present an acute circulatory failure for whom the physician in charge will decide to start a fluid expansion.

Hemodynamic variables will be obtained through transpulmonary thermodilution and pulse contour analysis (PICCO2 device, Pulsion Germany).

Fluid expansion will consist in the infusion of 500 ml of saline through a central venous catheter in a standardized 10-minutes period. The duration of infusion will be controlled by an airbag pressurized at 300 mmHg.

Fluid responsiveness will be defined by an increase in cardiac output over 15-per-cent from baseline (before fluid expansion).

Study design:

At time of decision to make the fluid expansion, a calibration of the PICCO2 device will be performed and a first set of hemodynamic measurements will be collected (cardiac output, cardiac function index, extravascular lung water, permeability vascular pulmonary index, global end diastolic volume, arterial pressure, heart rate).

Then, fluid expansion will be administrated in less than 10 minutes. From the start of fluid expansion to the end of the two-hours period ot time, pulse contour cardiac output and arterial pressure will be continuously recorded.

During the whole two hours period, no change in vasopressor dosage nor mechanical ventilation settings will be allowed.

In case of hemodynamic instability, defined by a mean arterial pressure under 65mmHg, a new fluid expansion could be realized. In this last case, the protocol will start again from the beginning.

ELIGIBILITY:
Inclusion Criteria:

* acute circulatory failure (infusion of norepinephrine)
* invasive mechanical ventilation through an endotracheal tube
* decision of fluid expansion

Non inclusion Criteria:

* extracorporeal membranous oxygenation (ECMO)
* active bleeding
* continuous renal replacement therapy with weight loss
* administration of diuretics within the past six hours
* decision of therapeutic limitation,
* age under eighteen years

Exclusion criteria:

* hemodynamic instability after fluid expansion (mean arterial pressure < 65mmHg)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted in the intensive care unit receiving mechanical ventilation and presenting an acute circulatory failure.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output during fluid expansion | 10 minutes
  Difference between maximal cardiac output during fluid expansion and baseline

SECONDARY OUTCOMES:
Change in cardiac output after fluid expansion | 2 hours
  Change in cardiac output after fluid expansion

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dres, MD, PhD, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nunes TS, Ladeira RT, Bafi AT, de Azevedo LC, Machado FR, Freitas FG. Duration of hemodynamic effects of crystalloids in patients with circulatory shock after initial resuscitation. Ann Intensive Care. 2014 Aug 1;4:25. doi: 10.1186/s13613-014-0025-9. eCollection 2014. PMID 25593742